CLINICAL TRIAL: NCT00725283
Title: Study of GSK2130579A Tumor-Antigen-Specific Cancer Immunotherapeutic as Post-consolidation Therapy in Adult Patients With Acute Myeloid Leukemia
Brief Title: Evaluation of a New Anti-cancer Immunotherapy After Chemotherapy in Adult Patients With Acute Myeloid Leukemia (AML)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 111444; 2010-023886-24 (EudraCT Number)
Record Dates: First submitted 2008-07-29; First posted 2008-07-30 (Estimated); Results first posted 2018-08-07 (Actual); Last update posted 2018-08-07 (Actual); Status verified 2017-06

CONDITIONS: Leukaemia, Myelocytic, Acute
Keywords: Leukemia; ASCI; Complete remission; Immunotherapy; adult; Acute Myeloid Leukemia; Tumor antigen; WT1
MeSH Terms: conditions — Leukemia; Pathologic Complete Response; Leukemia, Myeloid, Acute

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- GSK2130579A Group (Experimental): Patients with cytologically proven AML, as defined by the World Health Organization classification, who were administered a standard dose of GSK2130579A treatment. Patients received 24 doses of the study treatment over a period of approximately 4 years.
  Interventions: Biological: GSK Biologicals' recombinant WT1 Antigen-Specific Cancer Immunotherapeutic (ASCI)

INTERVENTIONS:
Biological: GSK Biologicals' recombinant WT1 Antigen-Specific Cancer Immunotherapeutic (ASCI) — Intramuscular administration
  Other Names: WT1 ASCI; GSK2130579A

SUMMARY:
This study is being done to evaluate the safety of a WT1 Antigen-Specific Cancer Immunotherapeutic (WT1 ASCI) as post-consolidation therapy in adult patients with WT1-positive Acute Myeloid Leukemia in first complete remission. It will also be analyzed to what extent this treatment induces an immune response, specific to the malignancy.

DETAILED DESCRIPTION:
In this study, patients were to receive a maximum of 24 doses of WT1 ASCI according four cycles over a period of four years.

This protocol summary has been updated according to the Protocol Amendment 6 (dated 10 Sept 2014).

There will no longer be an active follow-up of patients after discontinuation or completion of the treatment. The study will end 30 days after the last dose will be administered, so the patients will not be further exposed to unnecessary study related procedures.. In addition, no more biological samples will be collected for protocol research purposes. For each biological sample already collected in the scope of this study and not tested yet, testing will not be performed by default, except if a scientific rationale remains relevant. Blood sampling for safety monitoring as per protocol will continue.

ELIGIBILITY:
Inclusion Criteria:

* The patient has cytologically proven AML, as defined by the WHO classification. The pretreatment AML karyotype should be documented.
* The leukemia could be a de novo or secondary AML.
* The patient received induction and consolidation therapy according to the Institution's standard of care.
* The patient's blasts cells show expression of WT1 tran-script, detected by quantitative RT-PCR.
* The patient is in complete remission (i.e. CR1, CR2, …):
* Written informed consent has been obtained prior to the performance of any protocol-specific procedure.
* The patient is >= 18 years of age at the time of signature of the informed consent form.
* Eastern Cooperative Oncology Group performance status of 0, 1 or 2.
* Adequate hepatic and renal function defined as:

  * Serum bilirubin < 1.5 times the Upper Limit of Nor-mal (ULN).
  * Serum alanine aminotransferase < 2.5 times the ULN.
  * Calculated creatinine clearance > 50 mL/min.
* If the patient is female, she must be of non-childbearing potential, i.e. have a current tubal ligation, hysterectomy, ovariectomy or be post-menopausal, or if she is of childbearing potential, she must practice adequate con-traception for 30 days prior to treatment administration, have a negative pregnancy test and continue such pre-cautions for two months after completion of the treatment administration series.
* In the view of the investigator, the patient can and will comply with the requirements of the protocol.

Exclusion Criteria:

* The patient is in morphologic leukemia-free state or in morphologic complete remission with incomplete blood count recovery (CRi).
* The patient has acute promyelocytic leukemia with t(15;17)(q22;q12), (PML/RARα) or variants.
* The patient has received, or is receiving induction chemotherapy followed by Stem Cell Transplantation.
* The patient has (or has had) previous or concomitant malignancies, except effectively treated malignancy that is considered by the investigator highly likely to have been cured.
* The patient has hypercalcemia.
* The patient is known to be HIV-positive.
* The patient has symptomatic autoimmune disease such as, but not limited to multiple sclerosis, lupus, and in-flammatory bowel disease.
* The patient has a history of allergic reactions likely to be exacerbated by any component of the study investigational product.
* The patient has other concurrent severe medical prob-lems, unrelated to the malignancy, that would significantly limit full compliance with the study or expose the patient to unacceptable risk.
* The patient has a history of congestive heart failure, cor-onary artery disease or previous myocardial infarction.
* The patient has psychiatric or addictive disorders that may compromise his/her ability to give informed consent, or to comply with the study procedures.
* The patient has received any investigational or non-registered medicinal product other than the study medi-cation within 30 days preceding the first dose of study medication or plans to receive such a drug during the study period.
* The patient requires concomitant treatment with systemic corticosteroids or any other immunosuppressive agents. The use of prednisone, or equivalent, <0.5 mg/kg/day (absolute maximum 40 mg/day), or inhaled corticosteroids or topical steroids is permitted.
* The patient has received intravenous administration of antibiotics within 2 weeks prior to first study treatment or oral antibiotics within 1 week prior to first study treatment.
* For female patients: the patient is pregnant or lactating.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2008-10-01 (Actual); Primary Completion 2016-06-22 (Actual); Study Completion 2016-06-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (10):
- United States (9):
  - GSK Investigational Site, Tampa, Florida
  - GSK Investigational Site, Baltimore, Maryland
  - GSK Investigational Site, Worcester, Massachusetts
  - GSK Investigational Site, Buffalo, New York
  - GSK Investigational Site, New York, New York
  - GSK Investigational Site, Winston-Salem, North Carolina
  - GSK Investigational Site, Nashville, Tennessee
  - GSK Investigational Site, San Antonio, Texas
  - GSK Investigational Site, Seattle, Washington
- GSK Investigational Site, Grenoble, France

RESULTS

PARTICIPANT FLOW:
Groups:
- GSK2130579A Group: Patients with cytologically proven Acute Myeloid Leukemia (AML), as defined by the World Health Organization classification, who were administered a standard dose of GSK2130579A treatment. Patients received 24 doses of the study treatment over a period of approximately 4 years, administered in 4 cycles (Cycle 1: 6 doses, given at 2-week intervals; Cycle 2: 6 doses, given at 3-week intervals; Cycle 3: 4 doses, given at 6-week intervals; Cycle 4: 4 doses, given at 3-month intervals followed by other 4 doses, given at 6-month intervals).
Period: Overall Study
Arm/Group | GSK2130579A Group
Started | 34
Completed | 10
Not Completed | 24
Not completed — Missing Code | 3
Not completed — Death | 5
Not completed — Other | 6
Not completed — Withdrawal by Subject | 10

BASELINE CHARACTERISTICS:
Arm/Group | GSK2130579A Group
Number analyzed (Participants) | 34
Age, Continuous [Mean (Standard Deviation); unit: Years] | 60.1 (12.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18
  Male | 16
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With Severe Toxicities
Description: Severe toxicities (as classified according to the National Cancer Institute's Common Terminology Criteria for Adverse Events (CTCAE), Version 3.0) during the study treatment period defined as a study product-related or possibly study product-related:
  * Grade 4 toxicity (exception: Grade 4 fatigue - including lethargy, asthenia, and malaise - had to have a duration of at least 48 hours to be taken into account).
  * Grade 3 toxicity lasting for at least 48 hours (exceptions: myalgia, arthralgia, headache, and fever, regardless of duration).
  * An allergic reaction/hypersensitivity Grade 2 toxicity (i.e., rash, flushing, urticaria, and dyspnea). Drug fever was not part of this definition.
  * Decrease in renal function, with a calculated creatinine clearance < 40 mL/min.
  * Grade 2 cardiac ischemia/infarction (i.e., asymptomatic and testing suggesting ischemia; stable angina).
Time Frame: During the study treatment period (From Day 0 to Month 48)
Population: This analysis was performed on the Total treated population, which included all patients who had started treatment and received at least one dose of the study product, which were included in the overall safety analyses.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2130579A Group
Number analyzed (Participants) | 34
Participants
  Encephalitis | 1
  Rash erythematous | 1
  Hypersensitivity | 1
  Angina pectoris | 1
  Rash | 1
  Thrombocytopenia | 1

2. Primary Outcome: Seropositivity Rates for Anti-Wilms Tumor Antigen 1 (WT1) Antibodies
Description: Seropostivity rate was defined as the number of patients with anti-WT1 antibody concentration greater than or equal to (≥) the cut-off value of 9 Enzyme-linked Immunosorbent Assay (ELISA) units per milliliter (EU/mL).
Time Frame: At Baseline [Week 0], at Cycle 1 visits [Weeks 5, 9, 13], at Cycle 2 visits [Weeks 15, 21, 32], at Cycle 3 visits [Weeks 40, 54], at Cycle 4 visits [Months 15, 18, 21, 24, 30 and 49 (concluding visit)] and at Follow-up Visits [Months 52, 55, 58, 61]
Population: This analysis was performed on the Total treated population, which included all patients who had started treatment and received at least one dose of the study product, which were included in the overall safety analyses and for whom assay results were available at the considered timepoints.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2130579A Group
Number analyzed (Participants) | 31
Participants
  Week 0 | 2
  Week 5: number analyzed (Participants) | 27
  Week 5 | 6
  Week 9: number analyzed (Participants) | 23
  Week 9 | 21
  Week 13: number analyzed (Participants) | 24
  Week 13 | 24
  Week 15: number analyzed (Participants) | 21
  Week 15 | 21
  Week 21: number analyzed (Participants) | 21
  Week 21 | 21
  Week 32: number analyzed (Participants) | 19
  Week 32 | 19
  Week 40: number analyzed (Participants) | 18
  Week 40 | 18
  Week 54: number analyzed (Participants) | 16
  Week 54 | 16
  Month 15: number analyzed (Participants) | 12
  Month 15 | 12
  Month 18: number analyzed (Participants) | 9
  Month 18 | 9
  Month 21: number analyzed (Participants) | 6
  Month 21 | 6
  Month 24: number analyzed (Participants) | 5
  Month 24 | 5
  Month 30: number analyzed (Participants) | 1
  Month 30 | 1
  Month 49: number analyzed (Participants) | 20
  Month 49 | 15
  Month 52: number analyzed (Participants) | 11
  Month 52 | 7
  Month 55: number analyzed (Participants) | 12
  Month 55 | 7
  Month 58: number analyzed (Participants) | 7
  Month 58 | 6
  Month 61: number analyzed (Participants) | 3
  Month 61 | 3

3. Primary Outcome: Concentrations for Anti-WT1 Antibodies
Description: Antibody concentrations were presented as geometric mean concentrations (GMCs) and expressed as ELISA units per milliliter (EU/mL).
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: EU/mL
Arm/Group | GSK2130579A Group
Number analyzed (Participants) | 31
EU/mL
  Week 0 | 4.8 [4.4 to 5.2]
  Week 5: number analyzed (Participants) | 27
  Week 5 | 6.3 [4.8 to 8.3]
  Week 9: number analyzed (Participants) | 23
  Week 9 | 145.3 [66.3 to 318.5]
  Week 13: number analyzed (Participants) | 24
  Week 13 | 337.6 [185.2 to 615.4]
  Week 15: number analyzed (Participants) | 21
  Week 15 | 313.4 [165.0 to 595.4]
  Week 21: number analyzed (Participants) | 21
  Week 21 | 296.9 [162.2 to 543.5]
  Week 32: number analyzed (Participants) | 19
  Week 32 | 285.3 [165.3 to 492.4]
  Week 40: number analyzed (Participants) | 18
  Week 40 | 173.7 [100.7 to 299.8]
  Week 54: number analyzed (Participants) | 16
  Week 54 | 174.9 [103.0 to 296.8]
  Month 15: number analyzed (Participants) | 12
  Month 15 | 111.0 [53.5 to 230.0]
  Month 18: number analyzed (Participants) | 9
  Month 18 | 111.3 [41.5 to 298.3]
  Month 21: number analyzed (Participants) | 6
  Month 21 | 74.6 [22.3 to 249.5]
  Month 24: number analyzed (Participants) | 5
  Month 24 | 76.7 [12.8 to 459.3]
  Month 30: number analyzed (Participants) | 1
  Month 30 | 80.0 [NA to NA] — The lower and upper limits (LL and UL) of the confidence interval (CI) could not be configured due to only 1 participant at Month 30.
  Month 49: number analyzed (Participants) | 20
  Month 49 | 45.3 [19.6 to 105.0]
  Month 52: number analyzed (Participants) | 11
  Month 52 | 25.6 [9.6 to 68.5]
  Month 55: number analyzed (Participants) | 12
  Month 55 | 18.7 [8.3 to 42.1]
  Month 58: number analyzed (Participants) | 7
  Month 58 | 24.0 [11.9 to 48.6]
  Month 61: number analyzed (Participants) | 3
  Month 61 | 25.5 [14.2 to 45.8]

4. Primary Outcome: Number of Patients With Anti-WT1 Antibody Response
Description: Treatment response was defined as:
  For initially seronegative patients: post-administration antibody concentration ≥ 9 EU/ML; For initially seropositive patients: post-administration antibody concentration ≥ 2 fold the pre-vaccination antibody concentration.
Time Frame: At Cycle 1 visits [Weeks 5, 9, 13], at Cycle 2 visits [Weeks 15, 21, 32], at Cycle 3 visits [Weeks 40, 54], at Cycle 4 visits [Months 15, 18, 21, 24, 30 and 49 (concluding visit)] and at Follow-up Visits [Months 52, 55, 58, 61]
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2130579A Group
Number analyzed (Participants) | 25
Participants
  Week 5 | 4
  Week 9: number analyzed (Participants) | 21
  Week 9 | 20
  Week 13: number analyzed (Participants) | 22
  Week 13 | 22
  Week 15: number analyzed (Participants) | 19
  Week 15 | 19
  Week 21: number analyzed (Participants) | 19
  Week 21 | 19
  Week 32: number analyzed (Participants) | 17
  Week 32 | 17
  Week 40: number analyzed (Participants) | 16
  Week 40 | 16
  Week 54: number analyzed (Participants) | 14
  Week 54 | 14
  Month 15: number analyzed (Participants) | 10
  Month 15 | 10
  Month 18: number analyzed (Participants) | 7
  Month 18 | 7
  Month 21: number analyzed (Participants) | 4
  Month 21 | 4
  Month 24: number analyzed (Participants) | 3
  Month 24 | 3
  Month 30: number analyzed (Participants) | 1
  Month 30 | 1
  Month 49: number analyzed (Participants) | 20
  Month 49 | 15
  Month 52: number analyzed (Participants) | 11
  Month 52 | 7
  Month 55: number analyzed (Participants) | 12
  Month 55 | 7
  Month 58: number analyzed (Participants) | 7
  Month 58 | 6
  Month 61: number analyzed (Participants) | 3
  Month 61 | 3

5. Secondary Outcome: Number of Patients With Any Unsolicited Adverse Events
Description: An unsolicited AE covers any untoward medical occurrence in a clinical investigation subject temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product and reported in addition to those solicited during the clinical study and any solicited symptom with onset outside the specified period of follow-up for solicited symptoms. Any was defined as the occurrence of any unsolicited AE regardless of intensity grade or relation to vaccination.
Time Frame: Within the 31-day (Days 0-30) post-administration period
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2130579A Group
Number analyzed (Participants) | 34
Participants | 33

6. Secondary Outcome: Number of Patients With Any Serious Adverse Events (SAEs)
Description: Serious adverse events (SAEs) assessed include any medical occurrences that result in death, are life threatening, require hospitalization or prolongation of hospitalization or result in disability/incapacity. An event that was part of the natural course of the disease under study (i.e., disease progression, recurrence) was captured in the study as an efficacy measure, therefore, it did not need to be reported as an SAE. Death due to progressive disease was recorded on a specific form in the Clinical Report Form (CRF), but not as an SAE.
Time Frame: During the whole study duration (From Day 0 up to the concluding visit, at Month 49)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2130579A Group
Number analyzed (Participants) | 34
Participants | 8

7. Secondary Outcome: Number of Patients With Serious Adverse Events Related to Study Treatment
Description: Serious adverse events (SAEs) assessed include medical occurrences related to treatment administration that result in death, are life threatening, require hospitalization or prolongation of hospitalization or result in disability/incapacity. An event that was part of the natural course of the disease under study (i.e., disease progression, recurrence) was captured in the study as an efficacy measure, therefore, it did not need to be reported as an SAE. Death due to progressive disease was recorded on a specific form in the CRF, but not as an SAE.
Time Frame: During the whole study duration (From Day 0 up to the concluding visit, at Month 49)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2130579A Group
Number analyzed (Participants) | 34
Participants | 3

ADVERSE EVENTS:
Time Frame: Unsolicited adverse events (AEs): during the 31-day (Days 0-30) post-administration period; Serious adverse events (SAEs): during the entire study period (from Month 0 up to Month 49).
Arm/Group | GSK2130579A Group
All-Cause Mortality (participants affected / at risk) | 5/34
Serious Adverse Events (participants affected / at risk) | 8/34
Other Adverse Events (participants affected / at risk) | 33/34
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GSK2130579A Group (N=34)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1)
Myocardial infarction (Cardiac disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Oesophagitis (Gastrointestinal disorders) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1)
Hypersensitivity (Immune system disorders) | 1 (1)
Encephalitis (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 1 (2)
Upper respiratory tract infection (Infections and infestations) | 1 (1)
Viral infection (Infections and infestations) | 1 (1)
Wound infection (Infections and infestations) | 1 (1)
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GSK2130579A Group (N=34)
Anaemia (Blood and lymphatic system disorders) | 4 (5)
Increased tendency to bruise (Blood and lymphatic system disorders) | 2 (2)
Leukopenia (Blood and lymphatic system disorders) | 6 (6)
Lymphopenia (Blood and lymphatic system disorders) | 2 (2)
Neutropenia (Blood and lymphatic system disorders) | 6 (7)
Thrombocytopenia (Blood and lymphatic system disorders) | 10 (17)
Abdominal pain (Gastrointestinal disorders) | 5 (6)
Constipation (Gastrointestinal disorders) | 9 (10)
Diarrhoea (Gastrointestinal disorders) | 10 (15)
Dry mouth (Gastrointestinal disorders) | 2 (2)
Nausea (Gastrointestinal disorders) | 9 (24)
Vomiting (Gastrointestinal disorders) | 4 (7)
Asthenia (General disorders) | 4 (6)
Chills (General disorders) | 3 (4)
Cyst (General disorders) | 2 (2)
Fatigue (General disorders) | 17 (40)
Influenza like illness (General disorders) | 5 (6)
Injection site erythema (General disorders) | 5 (7)
Injection site pain (General disorders) | 22 (78)
Injection site pruritus (General disorders) | 4 (13)
Injection site reaction (General disorders) | 6 (15)
Injection site swelling (General disorders) | 3 (4)
Oedema peripheral (General disorders) | 6 (11)
Pain (General disorders) | 7 (9)
Pyrexia (General disorders) | 5 (6)
Bronchitis (Infections and infestations) | 3 (3)
Herpes zoster (Infections and infestations) | 3 (3)
Upper respiratory tract infection (Infections and infestations) | 10 (15)
Urinary tract infection (Infections and infestations) | 2 (3)
Contusion (Injury, poisoning and procedural complications) | 3 (3)
Procedural pain (Injury, poisoning and procedural complications) | 3 (4)
Skin abrasion (Injury, poisoning and procedural complications) | 2 (2)
Alanine aminotransferase increased (Investigations) | 2 (3)
Aspartate aminotransferase increased (Investigations) | 5 (6)
Decreased appetite (Metabolism and nutrition disorders) | 4 (5)
Hyperglycaemia (Metabolism and nutrition disorders) | 3 (5)
Hyperkalaemia (Metabolism and nutrition disorders) | 2 (3)
Hypokalaemia (Metabolism and nutrition disorders) | 4 (6)
Iron overload (Metabolism and nutrition disorders) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 6 (10)
Back pain (Musculoskeletal and connective tissue disorders) | 8 (9)
Bone pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 5 (5)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 2 (7)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 5 (6)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 2 (2)
Myalgia (Musculoskeletal and connective tissue disorders) | 4 (6)
Neck pain (Musculoskeletal and connective tissue disorders) | 3 (3)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 10 (19)
Dizziness (Nervous system disorders) | 16 (25)
Headache (Nervous system disorders) | 3 (3)
Hypoaesthesia (Nervous system disorders) | 2 (2)
Neuropathy peripheral (Nervous system disorders) | 2 (2)
Post herpetic neuralgia (Nervous system disorders) | 2 (2)
Sciatica (Nervous system disorders) | 2 (2)
Anxiety (Psychiatric disorders) | 4 (6)
Insomnia (Psychiatric disorders) | 5 (6)
Haematuria (Renal and urinary disorders) | 3 (3)
Breast pain (Reproductive system and breast disorders) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 5 (7)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 6 (7)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 2 (3)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 2 (3)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 2 (4)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 5 (9)
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 2 (3)
Dry skin (Skin and subcutaneous tissue disorders) | 6 (7)
Erythema (Skin and subcutaneous tissue disorders) | 5 (8)
Night sweats (Skin and subcutaneous tissue disorders) | 2 (2)
Onychoclasis (Skin and subcutaneous tissue disorders) | 2 (4)
Pruritus (Skin and subcutaneous tissue disorders) | 6 (9)
Rash (Skin and subcutaneous tissue disorders) | 5 (5)
Rash erythematous (Skin and subcutaneous tissue disorders) | 3 (5)
Skin lesion (Skin and subcutaneous tissue disorders) | 2 (2)
Hypertension (Vascular disorders) | 3 (3)
Hypotension (Vascular disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.